CLINICAL TRIAL: NCT05515523
Title: Pilot Trial of Intra-articular Stromal Vascular Fraction for the Treatment of Knee Post-Trauma Osteoarthritis and Biomarker Identification
Brief Title: Stromal Vascular Fraction (SVF) for Knee Post-Trauma Osteoarthritis (PTOA)
Acronym: SVF
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00088231
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis
Keywords: degenerative joint disease; degenerative arthritis; Knee trauma
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Intervention Model Description: single injection of autologous Adipose Derived (AD) Stromal Vascular Fraction (SVF) for the treatment of knee Post Traumatic Osteoarthritis (PTOA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- a single injection of autologous Adipose Derived (AD) Stromal Vascular Fraction (SVF) (Experimental): a single injection of autologous Adipose Derived (AD) Stromal Vascular Fraction (SVF) for the treatment of knee Post Traumatic Osteoarthritis (PTOA)
  Interventions: Genetic: Adipose Derived (AD) Stromal Vascular Fraction (SVF)

INTERVENTIONS:
Genetic: Adipose Derived (AD) Stromal Vascular Fraction (SVF) — autologous stromal vascular fraction cells from adipose tissue for reintroduction to the same patient during a single surgical procedure for treatment of pain and function associated with OA of the knee joint

SUMMARY:
This is a prospective, non-randomized, interventional, dual site, before-after clinical trial to determine feasibility and safety of a single injection of autologous Adipose Derived (AD) Stromal Vascular Fraction (SVF) for the treatment of knee Post Traumatic Osteoarthritis (PTOA).

DETAILED DESCRIPTION:
Clinical treatment generally involves a life-long combination of exercise, lifestyle modifications, and/or analgesics. If pain becomes debilitating, different surgical options exist, including arthroscopic joint debridement and mechanical axis change through osteotomies around the knee and eventually joint replacement surgery for severe cases to improve the quality of life. However, patients under 40 years of age, who expect to continue an active lifestyle, have only a 40% "good or excellent" function score after total knee replacement, they are most likely to outlive their initial replacement and need revision.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 45 with a preceding history (>1 and < 20 years ago) of significant knee trauma or trauma- related knee surgery
* Post-Trauma Osteoarthritis (PTOA) as diagnosed by K-L Grade II or III OA (weight bearing X-ray) and physician review
* Subjects must present with symptomatic (injured knee) visual analog scale (VAS) pain > 4. If bilateral disease, Knee Osteoarthritis (KOA) pain in the other knee must be less than/equal to 3 on the VAS for pain
* Subjects must have an adjusted Western Ontario and McMaster Universities Arthritis Index (WOMAC) (100-point scale) of > 25 and <90
* Study Subjects must have continued knee pain despite at least two conservative prescribed therapies (pain medications, physical therapy, knee injections, or weight loss), spanning a period of at least 3 months
* Study Subjects must be willing to voluntarily give written Informed Consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed
* Subjects will be in good health (ASA Class I-II) with a Body mass index (BMI) < 35
* Subjects must speak, read, and understand English
* Subjects must be reasonably able to return for multiple follow-up visits, to include procedure visits

Exclusion Criteria:

* Subjects whose knee pain is caused by, (i) diffuse edema, (ii) cartilage lesion greater than 1 cm width and grade 4 depth by MRI or (iii) osteochondritis dissecans
* Subjects who have had surgery of either knee within 12 months prior to the screening visit
* Subjects who have had an injection in either knee in the prior 3 months, including corticosteroids, viscosupplementation, stem cells, or platelet rich plasma (PRP)
* Subjects who have gout, rheumatoid arthritis, lupus arthropathy, psoriatic arthritis, avascular necrosis, severe bone deformity, infection of the knee joint, fibromyalgia, or neurogenic or vascular claudication
* Subjects who have symptomatic Osteoarthritis (OA) of the hips, spine, or ankle that would interfere with the evaluation of the treated knee
* Subjects that are unwilling to stop taking prescription or over the counter pain and anti-inflammatory medication for 7 days prior to any visit
* Subjects that are allergic to lidocaine, epinephrine, or valium or other sedatives
* Subjects with a history of bleeding disorders, anticoagulation therapy that cannot be stopped prior to IA injection
* Subjects with systemic immunosuppressant use within six (6) weeks from screening
* Subjects with human immunodeficiency virus (HIV)/viral hepatitis B or human T-lymphotropic virus type 1 (C/HTLV)
* Subjects with chondrocalcinosis, Paget's disease and Villonodular synovitis
* Subjects that use any form of tobacco
* Women that are pregnant or planning to become pregnant during the study
* Subjects on long term use of oral steroids or disease-modifying anti-rheumatic drugs
* History of any chemotherapy or radiation therapy of the targeted/treatment leg or adipose harvest site
* Subjects currently on worker's compensation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | Year 1
  number of safety events post injection

OTHER OUTCOMES:
Knee Pain scores - Visual Analog Scale (VAS) | Baseline, Month 1, Month 3, Month 6, and Year 1
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity
Knee Pain scores - The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, Month 1, Month 3, Month 6, and Year 1
  The WOMAC Pain score ranges from 0 to 20 with higher scores equating to greater pain with activities of daily living
Synovial Fluid Inflammatory Biomarker measurements | Baseline, Month 1, Month 3, Month 6, and Year 1
  Biomarkers will be measured before and after SVF treatment, and their relationships to post-trauma knee pain and function examined - Spearman correlation (measures the degree of association between two variables) will be used between changes in VAS or WOMAC score and changes in the eight biomarkers: (cluster of differentiation 14 (CD14), high-affinity receptor of human hemoglobin-haptoglobin complexes (CD163), Matrix metalloproteinase-3 (MMP-3), Vascular endothelial growth factor (VEGF), metallopeptidase inhibitor 1 (TIMP-1), Monocyte chemoattractant protein-1 (MCP-1), Soluble Vascular Cell Adhesion Molecule-1 (sVCAM-1) and Soluble intercellular adhesion molecule-1 (sICAM-1)
General Health scores - Patient-Reported Outcomes Measurement Information System (PROMIS 29) | Baseline, Month 1, Month 3, Month 6, and Year 1
  There is no total score, but each axis forms its own score. PROMIS assessments use an Item Response Theory (IRT) based score called Expected A Posteriori (EAP) scores, which are then transformed onto a final T-score metric - profile measure assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items for each domain

CONTACTS AND LOCATIONS:
Overall Officials: Claude T Moorman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No